CLINICAL TRIAL: NCT00418522
Title: A Six Month, Open Label, Randomized Parallel Group Trial Assessing The Impact Of Dry Powder Inhaled Insulin (Exubera) On Glycemic Control Compared To Insulin Glargine (Lantus) In Patients With Type 2 Diabetes Mellitus Who Are Poorly Controlled On A Combination Of Two Or More Oral Agents
Brief Title: This Study Is To Determine If Inhaled Insulin Is Effective In Treating Type 2 Diabetes Mellitus
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: A2171095
Record Dates: First submitted 2007-01-03; First posted 2007-01-05 (Estimated); Results first posted 2009-09-04 (Estimated); Last update posted 2018-09-28 (Actual); Status verified 2018-08

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: Insulin Glargine Diabetes HbA1c
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Insulin Glargine; Exubera

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Insulin glargine (Active Comparator): Insulin glargine, label instruction initiation dose (10 units), and individually adjusted doses, per subject's blood glucose, over the six months study, in addition to oral agents.
  Interventions: Drug: Insulin glargine
- Exubera (Experimental): Initiation dose of one mg per meal, and individually adjusted doses, per subject's blood glucose, over the six months study, in addition to oral agents.
  Interventions: Drug: Inhaled Insulin (Exubera)

INTERVENTIONS:
Drug: Insulin glargine — Insulin glargine, label instruction initiation dose (10 units), and individually adjusted doses, per subject's blood glucose, over the six months study, in addition to oral agents.
  Arms: Insulin glargine
Drug: Inhaled Insulin (Exubera) — Initiation dose of one mg per meal, and individually adjusted doses, per subject's blood glucose, over the six months study, in addition to oral agents.
  Arms: Exubera

SUMMARY:
This study is to determine if inhaled insulin is effective in treating type 2 diabetes mellitus.

ELIGIBILITY:
Inclusion Criteria:

* Age > 30 years and ≤ 75 years with a diagnosis of type 2 diabetes mellitus made > 6 months prior to study entry
* Screening HbA1c > 7.0%
* Currently treated on a stable dose of at least 2 oral antidiabetic agents for at least 3 months prior to study entry; including a sulfonylurea and/or metformin, and/or a thiazolidinedione

Exclusion Criteria:

Smoking within last 6 months PFTs outside of range

* Type 1 diabetes mellitus
* Type 2 diabetes mellitus currently (last three months) treated with an insulin regimen (alone or with Oral Antidiabetic Agents)
* Active liver disease; significantly-impaired hepatic function, as shown by, but not limited to, alanine aminotransferase (ALT) serum glutamic pyruvic transaminase (SGPT) or aspartate transaminase (AST) serum glutamic-oxaloacetic transaminase (SGOT) above 2x the upper limit of normal as measured at visit 1. However, patients with elevated ALT >1.5 upper limit of normal as a result of hepatic steatosis are permitted to enter the study.

Ages: 30 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 413 (Actual)
Dates: Start 2007-03; Primary Completion 2008-08 (Actual); Study Completion 2008-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (67):
- United States (66):
  - Pfizer Investigational Site, Phoenix, Arizona
  - Pfizer Investigational Site, Tucson, Arizona
  - Pfizer Investigational Site, Concord, California
  - Pfizer Investigational Site, Encino, California
  - Pfizer Investigational Site, Fresno, California
  - Pfizer Investigational Site, Fullerton, California
  - Pfizer Investigational Site, Long Beach, California
  - Pfizer Investigational Site, Mission Viejo, California
  - Pfizer Investigational Site, Pasadena, California
  - Pfizer Investigational Site, San Diego, California
  - Pfizer Investigational Site, San Luis Obispo, California
  - Pfizer Investigational Site, Spring Valley, California
  - Pfizer Investigational Site, Stockton, California
  - Pfizer Investigational Site, Walnut Creek, California
  - Pfizer Investigational Site, West Hills, California
  - Pfizer Investigational Site, Golden, Colorado
  - Pfizer Investigational Site, Waterbury, Connecticut
  - Pfizer Investigational Site, Newark, Delaware
  - Pfizer Investigational Site, Chiefland, Florida
  - Pfizer Investigational Site, Clearwater, Florida
  - Pfizer Investigational Site, Hollywood, Florida
  - Pfizer Investigational Site, Kissimmee, Florida
  - Pfizer Investigational Site, Miami, Florida
  - Pfizer Investigational Site, Ocala, Florida
  - Pfizer Investigational Site, Saint Cloud, Florida
  - Pfizer Investigational Site, Winter Park, Florida
  - Pfizer Investigational Site, Atlanta, Georgia
  - Pfizer Investigational Site, Lawrenceville, Georgia
  - Pfizer Investigational Site, Woodstock, Georgia
  - Pfizer Investigational Site, Boise, Idaho
  - Pfizer Investigational Site, Hayden Lake, Idaho
  - Pfizer Investigational Site, Indianapolis, Indiana
  - Pfizer Investigational Site, Overland Park, Kansas
  - Pfizer Investigational Site, Topeka, Kansas
  - Pfizer Investigational Site, Lexington, Kentucky
  - Pfizer Investigational Site, Louisville, Kentucky
  - Pfizer Investigational Site, Baton Rouge, Louisiana
  - Pfizer Investigational Site, New Orleans, Louisiana
  - Pfizer Investigational Site, Haverhill, Massachusetts
  - Pfizer Investigational Site, Springfield, Missouri
  - Pfizer Investigational Site, Omaha, Nebraska
  - Pfizer Investigational Site, Las Vegas, Nevada
  - Pfizer Investigational Site, Staten Island, New York
  - Pfizer Investigational Site, Charlotte, North Carolina
  - Pfizer Investigational Site, Statesville, North Carolina
  - Pfizer Investigational Site, Winston-Salem, North Carolina
  - Pfizer Investigational Site, Kettering, Ohio
  - Pfizer Investigational Site, Maumee, Ohio
  - Pfizer Investigational Site, Toledo, Ohio
  - Pfizer Investigational Site, Oklahoma City, Oklahoma
  - Pfizer Investigational Site, Medford, Oregon
  - Pfizer Investigational Site, Melrose Park, Pennsylvania
  - Pfizer Investigational Site, Greenville, South Carolina
  - Pfizer Investigational Site, Greer, South Carolina
  - Pfizer Investigational Site, Spartanburg, South Carolina
  - Pfizer Investigational Site, Milan, Tennessee
  - Pfizer Investigational Site, Arlington, Texas
  - Pfizer Investigational Site, Beaumont, Texas
  - Pfizer Investigational Site, Dallas, Texas
  - Pfizer Investigational Site, El Paso, Texas
  - Pfizer Investigational Site, Houston, Texas
  - Pfizer Investigational Site, San Antonio, Texas
  - Pfizer Investigational Site, Bennington, Vermont
  - Pfizer Investigational Site, Richmond, Virginia
  - Pfizer Investigational Site, Federal Way, Washington
  - Pfizer Investigational Site, Menomonee Falls, Wisconsin
- Pfizer Investigational Site, Carolina, Puerto Rico

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A2171095&StudyName=This%20Study%20Is%20To%20Determine%20If%20Inhaled%20Insulin%20Is%20Effective%20In%20Treating%20Type%202%20Diabetes%20Mellitus

RESULTS

PARTICIPANT FLOW:
Groups:
- Inhaled Human Insulin: Initiation dose of 1 milligram per meal, and individually adjusted doses, per subject's blood glucose, over the 6 month study, in addition to oral agents.
Period: Overall Study
Arm/Group | Inhaled Human Insulin | Insulin Glargine
Started | 219 | 194
Received Treatment | 212 | 190
Completed | 136 | 152
Not Completed | 83 | 42
Not completed — Adverse Event | 7 | 1
Not completed — Lack of Efficacy | 1 | 3
Not completed — Lost to Follow-up | 10 | 4
Not completed — Withdrawal by Subject | 31 | 7
Not completed — Other | 27 | 23
Not completed — Randomized but did not receive treatment | 7 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Inhaled Human Insulin | Insulin Glargine | Total
Number analyzed (Participants) | 212 | 190 | 402
Age, Customized [Number; unit: participants]
  18 to 44 years | 27 | 26 | 53
  45 to 65 years | 151 | 125 | 276
  >=65 years | 34 | 39 | 73
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 92 | 84 | 176
  Male | 120 | 106 | 226

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Glycosylated Hemoglobin A1c (HbA1c) at Week 26 for the Per Protocol (PP) Population
Description: HbA1c lab value: Change = value at Week 26 minus value at Baseline.
Time Frame: Baseline, Week 26
Population: Per protocol (PP)=Full Analysis Set (FAS) subjects (i.e., had >=1 study drug dose and >=1 post-baseline measurement) with >=12 weeks treatment and no major protocol violation. LOCF imputed missing data with any post-baseline visit. Number of subjects with HbA1c values at Baseline and Week 26: inhaled human insulin n=154, insulin glargine n=157.
Measure: Mean (Standard Deviation); unit: percent
Arm/Group | Inhaled Human Insulin | Insulin Glargine
Number analyzed (Participants) | 154 | 157
percent | -2.01 (1.39) | -1.75 (1.40)
Statistical Analysis 1: Comparison: Inhaled Human Insulin vs Insulin Glargine; The null hypothesis was that the inhaled human insulin group was inferior to the insulin glargine group with respect to 26-week change from baseline in HbA1c, while the alternate hypothesis is that the inhaled human insulin group was not inferior to the insulin glargine group with respect to 26-week change from baseline in HbA1c, given the predetermined non-inferiority margin of 0.4%; Test type: Non-Inferiority or Equivalence — The non-inferiority test utilized a one-sided 2.5% level of significance; p < 0.0001, ANCOVA; Mean Difference (Final Values) = -0.19, 95% CI [-0.38 to 0] — A confidence interval (CI) approach was presented with a two-sided 95% CI of the difference between treatment and control
Statistical Analysis 2: Comparison: Inhaled Human Insulin vs Insulin Glargine; With an established non-inferiority claim, an additional test for superiority was conducted (ie, the margin was 0.0%); Test type: Superiority or Other; p = 0.0516, ANCOVA; Mean Difference (Final Values) = -0.19, 95% CI [-0.38 to 0] — The superiority test used a one-sided 2.5% level of significance

2. Secondary Outcome: Percentage of Subjects Achieving Glycemic Control (HbA1c < 6.5%) at Week 26
Description: Percentage of subjects with glycosylated hemoglobin A1c lab value less than 6.5%.
Time Frame: Week 26
Population: FAS=all subjects who took at least 1 dose of study drug and had at least 1 post-baseline measurement. LOCF imputed missing data with any post-baseline visit. Number of subjects with HbA1c < 6.5% at Week 26: inhaled human insulin n=72, insulin glargine n=42.
Measure: Number; unit: percentage of participants
Arm/Group | Inhaled Human Insulin | Insulin Glargine
Number analyzed (Participants) | 203 | 189
percentage of participants | 35.5 | 22.2
Statistical Analysis 1: Comparison: Inhaled Human Insulin vs Insulin Glargine; Test type: Superiority or Other; p = 0.0052, Regression, Logistic; Odds Ratio (OR) = 1.96, 95% CI [1.22 to 3.14]

3. Secondary Outcome: Percentage of Subjects Achieving Glycemic Control (HbA1c < 7.0%) at Week 26
Description: Percentage of subjects with glycosylated hemoglobin A1c lab value less than 7.0%.
Time Frame: Week 26
Population: FAS=all subjects who took at least 1 dose of study drug and had at least 1 post-baseline measurement. LOCF imputed missing data with any post-baseline visit. Number of subjects with HbA1c < 7.0% at Week 26: inhaled human insulin n=127, insulin glargine n=90.
Measure: Number; unit: percentage of participants
Arm/Group | Inhaled Human Insulin | Insulin Glargine
Number analyzed (Participants) | 203 | 189
percentage of participants | 62.6 | 47.6
Statistical Analysis 1: Comparison: Inhaled Human Insulin vs Insulin Glargine; Test type: Superiority or Other; p = 0.0022, Regression, Logistic; Odds Ratio (OR) = 2.01, 95% CI [1.29 to 3.15]

4. Secondary Outcome: Percentage of Subjects Achieving Glycemic Control (HbA1c < 8.0%) at Week 26
Description: Number of subjects with glycosylated hemoglobin A1c lab value less than 8.0%.
Time Frame: Week 26
Population: FAS=all subjects who took at least 1 dose of study drug and had at least 1 post-baseline measurement. LOCF imputed missing data with any post-baseline visit. Number of subjects with HbA1c < 8.0% at Week 26: inhaled human insulin n=162, insulin glargine n=158.
Measure: Number; unit: percentage of participants
Arm/Group | Inhaled Human Insulin | Insulin Glargine
Number analyzed (Participants) | 203 | 189
percentage of participants | 79.8 | 83.6
Statistical Analysis 1: Comparison: Inhaled Human Insulin vs Insulin Glargine; Test type: Superiority or Other; p = 0.2480, Regression, Logistic; Odds Ratio (OR) = 0.71, 95% CI [0.40 to 1.27]

5. Secondary Outcome: Change From Baseline in Fasting Plasma Glucose at Week 26
Description: Fasting plasma glucose lab value: Change = value at Week 26 minus value at Baseline.
Time Frame: Baseline, Week 26
Population: FAS=all subjects who took at least 1 dose of study drug and had at least 1 post-baseline measurement. LOCF imputed missing data with any post-baseline visit. Number of subjects with fasting plasma glucose at Baseline and Week 26: inhaled human insulin n=202, insulin glargine n=189.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Inhaled Human Insulin | Insulin Glargine
Number analyzed (Participants) | 203 | 189
mg/dL | -52.77 (69.48) | -53.50 (62.92)
Statistical Analysis 1: Comparison: Inhaled Human Insulin vs Insulin Glargine; Test type: Superiority or Other; p = 0.6091, ANCOVA; Mean Difference (Final Values) = 2.57, 95% CI [-7.31 to 12.46]

6. Secondary Outcome: Change From Baseline in Fasting and Postprandial Blood Glucose as Determined by Standardized Meal Tolerance Tests at Week 26
Description: Postprandial blood glucose lab value (Time 0 min [fasting], Time 30 min, Time 60 min, Time 90 min, Time 120 min, Time 180 min): Change = value at Week 26 minus value at Baseline.
Time Frame: Baseline, Week 26
Population: FAS=all subjects who took at least 1 dose of study drug and had at least 1 post-baseline measurement. LOCF imputed missing data with any post-baseline visit. Number of subjects with fasting and postprandial blood glucose measurements determined by standardized meal tolerance tests at Baseline and Week 26: n=inhaled human insulin, insulin glargine.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Inhaled Human Insulin | Insulin Glargine
Number analyzed (Participants) | 203 | 189
mg/dL
  Time 0 at Week 26 (n=105, 119) | -35.22 (51.12) | -61.16 (54.68)
  Time 30 at Week 26 (n=95, 107) | -49.91 (62.41) | -66.02 (62.32)
  Time 60 at Week 26 (n=110, 118) | -56.83 (69.81) | -64.77 (64.47)
  Time 90 at Week 26 (n=114, 120) | -64.94 (75.67) | -58.85 (64.58)
  Time 120 at Week 26 (n=113, 124) | -66.59 (74.69) | -54.89 (63.02)
  Time 180 at Week 26 (n=114, 122) | -66.99 (74.19) | -51.27 (59.92)
Statistical Analysis 1: Comparison: Inhaled Human Insulin vs Insulin Glargine; Time 0 (fasting) at Week 26; Test type: Superiority or Other; p < 0.0001, ANCOVA; Mean Difference (Final Values) = 32.96, 95% CI [22.66 to 43.25]
Statistical Analysis 2: Comparison: Inhaled Human Insulin vs Insulin Glargine; Time 30 at Week 26; Test type: Superiority or Other; p < 0.0001, ANCOVA; Mean Difference (Final Values) = 28.57, 95% CI [16.55 to 40.59]
Statistical Analysis 3: Comparison: Inhaled Human Insulin vs Insulin Glargine; Time 60 at Week 26; Test type: Superiority or Other; p = 0.0044, ANCOVA; Mean Difference (Final Values) = 18.96, 95% CI [5.96 to 31.96]
Statistical Analysis 4: Comparison: Inhaled Human Insulin vs Insulin Glargine; Time 90 at Week 26; Test type: Superiority or Other; p = 0.3168, ANCOVA; Mean Difference (Final Values) = 6.69, 95% CI [-6.45 to 19.83]
Statistical Analysis 5: Comparison: Inhaled Human Insulin vs Insulin Glargine; Time 120 at Week 26; Test type: Superiority or Other; p = 0.9222, ANCOVA; Mean Difference (Final Values) = 0.63, 95% CI [-12.12 to 13.39]
Statistical Analysis 6: Comparison: Inhaled Human Insulin vs Insulin Glargine; Time 180 at Week 26; Test type: Superiority or Other; p = 0.6950, ANCOVA; Mean Difference (Final Values) = -2.41, 95% CI [-14.51 to 9.69]

7. Secondary Outcome: Change From Baseline in Postprandial Blood Glucose as Measured by 8-Point Profiles at Week 26
Description: Post-prandial=after a meal. 8-point scale: (1 = before breakfast, 2 = 2 hours post breakfast, 3 = before lunch, 4 = 2 hours post lunch, 5 = before dinner, 6 = 2 hours post dinner, 7 = at bedtime, 8 = overnight [between 2 and 4 am]). Postprandial blood glucose lab value: Change = value at Week 26 minus value at Baseline.
Time Frame: Baseline, Week 26
Population: FAS = all subjects who took at least 1 dose of study drug and had at least 1 post-baseline measurement. LOCF imputed missing data with any post-baseline visit. Number of subjects with postprandial blood glucose measurements as measured by 8-point profiles at Baseline and Week 26: n=inhaled human insulin, insulin glargine.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Inhaled Human Insulin | Insulin Glargine
Number analyzed (Participants) | 203 | 189
mg/dL
  Post-Breakfast, Week 26 (n=185,171) | -86.61 (85.98) | -75.36 (79.04)
  Post-Lunch, Week 26 (n=184, 172) | -86.66 (77.49) | -58.51 (86.93)
  Post-Dinner, Week 26 (n=187,166) | -81.86 (75.94) | -59.20 (86.21)
Statistical Analysis 1: Comparison: Inhaled Human Insulin vs Insulin Glargine; Post-Breakfast, Week 26; Test type: Superiority or Other; p = 0.1207, ANCOVA; Mean Difference (Final Values) = -9.61, 95% CI [-21.76 to 2.54]
Statistical Analysis 2: Comparison: Inhaled Human Insulin vs Insulin Glargine; Post-Lunch, Week 26; Test type: Superiority or Other; p < 0.0001, ANCOVA; Mean Difference (Final Values) = -29.11, 95% CI [-39.77 to -18.44]
Statistical Analysis 3: Comparison: Inhaled Human Insulin vs Insulin Glargine; Post-Dinner, Week 26; Test type: Superiority or Other; p < 0.0001, ANCOVA; Mean Difference (Final Values) = -33.76, 95% CI [-44.17 to -23.35]

8. Secondary Outcome: Change From Baseline in Lipids at Week 26
Description: Lipid (total cholesterol, high density lipoprotein cholesterol [HDL-c], low density lipoprotein cholesterol [LDL-c], triglycerides) lab value: Change = value at Week 26 minus value at Baseline.
Time Frame: Baseline, Week 26
Population: FAS=all subjects who took at least 1 dose of study drug and had at least 1 post-baseline measurement. LOCF imputed missing data with any post-baseline visit. Number of subjects with lipids data at Baseline and Week 26: n=inhaled human insulin, insulin glargine.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Inhaled Human Insulin | Insulin Glargine
Number analyzed (Participants) | 203 | 189
mg/dL
  Total cholesterol, Week 26 (n=197, 186) | -2.80 (31.97) | -6.19 (29.95)
  HDL-c, Week 26 (n=197, 186) | 2.97 (6.99) | 0.69 (6.07)
  LDL-c, Week 26 (n=197, 186) | -2.09 (25.74) | -3.71 (23.63)
  Triglycerides, Week 26 (n=197, 187) | -42.65 (87.70) | -46.23 (147.8)
Statistical Analysis 1: Comparison: Inhaled Human Insulin vs Insulin Glargine; Total Cholesterol at Week 26; Test type: Superiority or Other; p = 0.0735, ANCOVA; Mean Difference (Final Values) = 5.21, 95% CI [-0.50 to 10.91]
Statistical Analysis 2: Comparison: Inhaled Human Insulin vs Insulin Glargine; HDL-c at Week 26; Test type: Superiority or Other; p = 0.0017, ANCOVA; Mean Difference (Final Values) = 2.09, 95% CI [0.79 to 3.39]
Statistical Analysis 3: Comparison: Inhaled Human Insulin vs Insulin Glargine; LDL-c at Week 26; Test type: Superiority or Other; p = 0.1369, ANCOVA; Mean Difference (Final Values) = 3.43, 95% CI [-1.10 to 7.96]
Statistical Analysis 4: Comparison: Inhaled Human Insulin vs Insulin Glargine; Triglycerides at Week 26; Test type: Superiority or Other; p = 0.5684, ANCOVA; Mean Difference (Final Values) = 4.26, 95% CI [-10.40 to 18.92]

9. Secondary Outcome: Change From Baseline in Cardiovascular (CV) Biomarkers High Sensitivity C-reactive Protein (Hs-CRP), Leptin, and Spot Urine Microalbumin at Week 26
Description: CV biomarker (hs-CRP, Leptin, and Spot Urine Microalbumin) lab value: Change = value at Week 26 minus value at Baseline.
Time Frame: Baseline, Week 26
Population: FAS=all subjects who took at least 1 dose of study drug and had at least 1 post-baseline measurement. LOCF imputed missing data with any post-baseline visit. Number of subjects with CV biomarker data (hs-CRP, leptin, and spot urine microalbumin) at Baseline and Week 26: n=inhaled human insulin, insulin glargine.
Measure: Mean (Standard Deviation); unit: mg/L
Arm/Group | Inhaled Human Insulin | Insulin Glargine
Number analyzed (Participants) | 203 | 189
mg/L
  hs-CRP, Week 26 (n=198, 187) | 0.61 (4.56) | 0.32 (3.69)
  Leptin, Week 26 (n=193, 186) | 3.68 (13.50) | 4.41 (10.50)
  Spot Urine Microalbumin, Week 26 (n=183, 169) | 3.47 (96.48) | 3.70 (54.53)
Statistical Analysis 1: Comparison: Inhaled Human Insulin vs Insulin Glargine; hs-CRP at Week 26; Test type: Superiority or Other; p = 0.5673, ANCOVA; Mean Difference (Final Values) = 0.24, 95% CI [-0.58 to 1.06]
Statistical Analysis 2: Comparison: Inhaled Human Insulin vs Insulin Glargine; Leptin at Week 26; Test type: Superiority or Other; p = 0.6099, ANCOVA; Mean Difference (Final Values) = -0.61, 95% CI [-2.97 to 1.75]
Statistical Analysis 3: Comparison: Inhaled Human Insulin vs Insulin Glargine; Spot urine microalbumin at Week 26; Test type: Superiority or Other; p = 0.7684, ANCOVA; Mean Difference (Final Values) = 2.28, 95% CI [-12.94 to 17.51]

10. Secondary Outcome: Change From Baseline in CV Biomarkers Adiponectin and Apolipoprotein B (ApoB) at Week 26
Description: CV biomarker (adiponectin and ApoB) lab value: Change = value at Week 26 minus value at Baseline.
Time Frame: Baseline, Week 26
Population: FAS=all subjects who took at least 1 dose of study drug and had at least 1 post-baseline measurement. LOCF imputed missing data with any post-baseline visit. Number of subjects with CV biomarker data (adiponectin and ApoB) at Baseline and Week 26: n=inhaled human insulin, insulin glargine.
Measure: Mean (Standard Deviation); unit: mg/mL
Arm/Group | Inhaled Human Insulin | Insulin Glargine
Number analyzed (Participants) | 203 | 189
mg/mL
  Adiponectin, Week 26 (n=195, 184) | 0.23 (5.58) | -0.32 (5.15)
  ApoB, Week 26 (n=198, 187) | -0.06 (0.19) | -0.06 (0.17)
Statistical Analysis 1: Comparison: Inhaled Human Insulin vs Insulin Glargine; Adiponectin at Week 26; Test type: Superiority or Other; p = 0.5005, ANCOVA; Mean Difference (Final Values) = 0.36, 95% CI [-0.69 to 1.42]
Statistical Analysis 2: Comparison: Inhaled Human Insulin vs Insulin Glargine; ApoB at Week 26; Test type: Superiority or Other; p = 0.6850, ANCOVA; Mean Difference (Final Values) = 0.01, 95% CI [-0.03 to 0.04]

11. Secondary Outcome: Change From Baseline in 24-Hour Continuous Glucose Monitoring System (CGMS) Glucose Values at Week 26
Description: 24-Hour CGMS glucose lab value was obtained using the Medtronic MiniMed CGMS. Not all subjects were offered the opportunity to participate in this assessment. Change = value at Week 26 minus value at Baseline.
Time Frame: Baseline, Week 26
Population: FAS-CGMS=all subjects with at least 1 study drug dose, at least 1 post-baseline measurement, and who participated in a 24-hour CGMS substudy. LOCF imputed missing data with any post-baseline visit. Number of subjects who participated in the substudy with 24-hour CGMS values at Baseline and Week 26: inhaled human insulin n=2, insulin glargine n=8.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Inhaled Human Insulin | Insulin Glargine
Number analyzed (Participants) | 203 | 189
mg/dL | -36.53 (33.96) | -35.63 (58.19)
Statistical Analysis 1: Comparison: Inhaled Human Insulin vs Insulin Glargine; Test type: Superiority or Other; p = 0.1856, ANCOVA; Mean Difference (Final Values) = 58.70, 95% CI [-43.37 to 160.77]

12. Secondary Outcome: Change From Baseline in Mean Standard Deviation (SD) of 24-Hour Glucose Values Measured by CGMS at Week 26
Description: SD of 24-Hour CGMS glucose lab value obtained using the Medtronic MiniMed CGMS. Not all subjects were offered the opportunity to participate in this assessment. Change = value at Week 26 minus value at Baseline.
Time Frame: Baseline, Week 26
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Inhaled Human Insulin | Insulin Glargine
Number analyzed (Participants) | 203 | 189
mg/dL | -12.50 (2.55) | 4.46 (11.51)
Statistical Analysis 1: Comparison: Inhaled Human Insulin vs Insulin Glargine; Test type: Superiority or Other; p = 0.1862, ANCOVA; Mean Difference (Final Values) = -18.72, 95% CI [-51.34 to 13.89]

13. Secondary Outcome: Number of Subjects With Hypoglycemic Events
Description: A hypoglycemic event was identified by characteristic symptoms or blood glucose levels. An event was severe if the subject was unable to treat him/herself; had at least 1 neurological symptom; or blood glucose of < = 49 mg/dL. Events not meeting all 3 criteria were considered mild-moderate. Overall=mild, moderate, and severe.
Time Frame: Months 1 to 7
Population: Safety population=all subjects who took at least 1 dose of study drug. Number of subjects with at least 1 hypoglycemic event during the course of the study that were evaluable at the specified month: n=inhaled human insulin, insulin glargine.
Measure: Number; unit: participants
Arm/Group | Inhaled Human Insulin | Insulin Glargine
Number analyzed (Participants) | 212 | 190
participants
  Overall at Month 1 (n=147, 83) | 70 | 24
  Mild/Moderate at Month 1 (n=147, 83) | 69 | 24
  Severe at Month 1 (n=147, 83) | 0 | 0
  Overall at Month 2 (n=141, 81) | 98 | 38
  Mild/Moderate at Month 2 (n=141, 81) | 98 | 38
  Severe at Month 2 (n=141, 81) | 1 | 0
  Overall at Month 3 (n=135, 81) | 84 | 35
  Mild/Moderate at Month 3 (n=135, 81) | 83 | 35
  Severe at Month 3 (n=135, 81) | 3 | 0
  Overall at Month 4 (n=120, 80) | 61 | 25
  Mild/Moderate at Month 4 (n=120, 80) | 61 | 25
  Severe at Month 4 (n=120, 80) | 0 | 0
  Overall at Month 5 (n=117, 79) | 55 | 30
  Mild/Moderate at Month 5 (n=117, 79) | 55 | 30
  Severe at Month 5 (n=117, 79) | 0 | 0
  Overall at Month 6 (n=109, 77) | 42 | 31
  Mild/Moderate at Month 6 (n=109, 77) | 42 | 31
  Severe at Month 6 (n=109, 77) | 0 | 0
  Overall at Month 7 (n=77, 60) | 8 | 4
  Mild/Moderate at Month 7 (n=77, 60) | 8 | 4
  Severe at Month 7 (n=77, 60) | 0 | 0

14. Secondary Outcome: Number of Total Hypoglycemic Events
Description: A hypoglycemic event was identified by characteristic symptoms or blood glucose levels. Severe=the subject was unable to treat him/herself; had at least 1 neurological symptom; or blood glucose of < = 49 mg/dL. Events not meeting all 3 criteria were considered mild-moderate. Overall=mild, moderate, and severe. Total=events during the study.
Time Frame: Months 1 to 7
Population: as for outcome 13
Measure: Number; unit: events
Arm/Group | Inhaled Human Insulin | Insulin Glargine
Number analyzed (Participants) | 212 | 190
events
  Overall at Month 1 (n=147, 83) | 195 | 41
  Mild/Moderate at Month 1 (n=147, 83) | 194 | 41
  Severe at Month 1 (n=147, 83) | 0 | 0
  Overall at Month 2 (n=141, 81) | 365 | 66
  Mild/Moderate at Month 2 (n=141, 81) | 364 | 66
  Severe at Month 2 (n=141, 81) | 1 | 0
  Overall at Month 3 (n=135, 81) | 292 | 84
  Mild/Moderate at Month 3 (n=135, 81) | 289 | 84
  Severe at Month 3 (n=135, 81) | 3 | 0
  Overall at Month 4 (n=120, 80) | 166 | 51
  Mild/Moderate at Month 4 (n=120, 80) | 166 | 51
  Severe at Month 4 (n=120, 80) | 0 | 0
  Overall at Month 5 (n=117, 79) | 157 | 64
  Mild/Moderate at Month 5 (n=117, 79) | 157 | 64
  Severe at Month 5 (n=117, 79) | 0 | 0
  Overall at Month 6 (n=109, 77) | 119 | 63
  Mild/Moderate at Month 6 (n=109, 77) | 119 | 63
  Severe at Month 6 (n=109, 77) | 0 | 0
  Overall at Month 7 (n=77, 60) | 12 | 5
  Mild/Moderate at Month 7 (n=77, 60) | 12 | 5
  Severe at Month 7 (n=77, 60) | 0 | 0

15. Secondary Outcome: Number of Total Subject Months of Treatment
Description: Number of total subject months of treatment. Subject months = number of days from start of treatment to the last day of active treatment + 1 day lag, including off-drug time)/30.44. Severe=the subject was unable to treat him/herself; had at least 1 neurological symptom; or blood glucose of < = 49 mg/dL. Events not meeting all 3 criteria were considered mild-moderate. Overall=mild, moderate, and severe.
Time Frame: Months 1 to 7
Population: as for outcome 13
Measure: Number; unit: subject months
Arm/Group | Inhaled Human Insulin | Insulin Glargine
Number analyzed (Participants) | 212 | 190
subject months
  Overall at Month 1 (n=147, 83) | 145.8 | 82.4
  Mild/Moderate at Month 1 (n=147, 83) | 145.8 | 82.4
  Severe at Month 1 (n=147, 83) | 145.8 | 82.4
  Overall at Month 2 (n=141, 81) | 138.3 | 81.0
  Mild/Moderate at Month 2 (n=141, 81) | 138.3 | 81.0
  Severe at Month 2 (n=141, 81) | 138.3 | 81.0
  Overall at Month 3 (n=135, 81) | 128.8 | 80.4
  Mild/Moderate at Month 3 (n=135, 81) | 128.8 | 80.4
  Severe at Month 3 (n=135, 81) | 128.8 | 80.4
  Overall at Month 4 (n=120, 80) | 117.7 | 79.7
  Mild/Moderate at Month 4 (n=120, 80) | 117.7 | 79.7
  Severe at Month 4 (n=120, 80) | 117.7 | 79.7
  Overall at Month 5 (n=117, 79) | 112.2 | 77.9
  Mild/Moderate at Month 5 (n=117, 79) | 112.2 | 77.9
  Severe at Month 5 (n=117, 79) | 112.2 | 77.9
  Overall at Month 6 (n=109, 77) | 103.5 | 75.7
  Mild/Moderate at Month 6 (n=109, 77) | 103.5 | 75.7
  Severe at Month 6 (n=109, 77) | 103.5 | 75.7
  Overall at Month 7 (n=77, 60) | 12.8 | 6.6
  Mild/Moderate at Month 7 (n=77, 60) | 12.8 | 6.6
  Severe at Month 7 (n=77, 60) | 12.8 | 6.6

16. Secondary Outcome: Crude Hypoglycemic Event Rate
Description: crude event rate=(events)/(subject-months). Severe=the subject was unable to treat him/herself; had at least 1 neurological symptom; or blood glucose of < = 49 mg/dL. Events not meeting all 3 criteria were considered mild-moderate. Overall=mild, moderate, and severe.
Time Frame: Months 1 to 7
Population: as for outcome 13
Measure: Number; unit: events / subject-months
Arm/Group | Inhaled Human Insulin | Insulin Glargine
Number analyzed (Participants) | 212 | 190
events / subject-months
  Overall at Month 1 (n=147, 83) | 1.3 | 0.5
  Mild/Moderate at Month 1 (n=147, 83) | 1.3 | 0.5
  Severe at Month 1 (n=147, 83) | 0 | 0
  Overall at Month 2 (n=141, 81) | 2.6 | 0.8
  Mild/Moderate at Month 2 (n=141, 81) | 2.6 | 0.8
  Severe at Month 2 (n=141, 81) | 0.7 | 0
  Overall at Month 3 (n=135, 81) | 2.3 | 1.0
  Mild/Moderate at Month 3 (n=135, 81) | 2.2 | 1.0
  Severe at Month 3 (n=135, 81) | 2.3 | 0
  Overall at Month 4 (n=120, 80) | 1.4 | 0.6
  Mild/Moderate at Month 4 (n=120, 80) | 1.4 | 0.6
  Severe at Month 4 (n=120, 80) | 0 | 0
  Overall at Month 5 (n=117, 79) | 1.4 | 0.8
  Mild/Moderate at Month 5 (n=117, 79) | 1.4 | 0.8
  Severe at Month 5 (n=117, 79) | 0 | 0
  Overall at Month 6 (n=109, 77) | 1.2 | 0.8
  Mild/Moderate at Month 6 (n=109, 77) | 1.2 | 0.8
  Severe at Month 6 (n=109, 77) | 0 | 0
  Overall at Month 7 (n=77, 60) | 0.9 | 0.8
  Mild/Moderate at Month 7 (n=77, 60) | 0.9 | 0.8
  Severe at Month 7 (n=77, 60) | 0 | 0

17. Secondary Outcome: Number of Nocturnal Hypoglycemic Events
Description: A hypoglycemic event was identified by characteristic symptoms or blood glucose levels. Severe=the subject was unable to treat him/herself; had at least 1 neurological symptom; or blood glucose of < = 49 mg/dL. Events not meeting all 3 criteria were considered mild-moderate. Nocturnal hypoglycemia=event occuring from midnight to 5:59 am.
Time Frame: Months 1 to 7
Population: Safety population=all subjects who took at least 1 dose of study drug.
Measure: Number; unit: events
Arm/Group | Inhaled Human Insulin | Insulin Glargine
Number analyzed (Participants) | 212 | 190
events | 187 | 114

18. Secondary Outcome: Change From Baseline in Body Weight at Week 26
Description: Body weight value: Change = value at Week 26 minus value at Baseline.
Time Frame: Baseline, Week 26
Population: FAS=all subjects who took at least 1 dose of study drug and had at least 1 post-baseline measurement. LOCF imputed missing data with any post-baseline visit. Number of subjects with body weight measurements at Baseline and Week 26: inhaled human insulin n=192, insulin glargine n=183.
Measure: Mean (Standard Deviation); unit: kg
Arm/Group | Inhaled Human Insulin | Insulin Glargine
Number analyzed (Participants) | 203 | 189
kg | 3.55 (4.74) | 2.33 (3.80)
Statistical Analysis 1: Comparison: Inhaled Human Insulin vs Insulin Glargine; Test type: Superiority or Other; p = 0.0055, ANCOVA; Mean Difference (Final Values) = 1.20, 95% CI [0.35 to 2.04]

19. Secondary Outcome: Change From Baseline in Body Mass Index (BMI) at Week 26
Description: BMI value (kg/m2): Change = value at Week 26 minus value at Baseline.
Time Frame: Baseline, Week 26
Population: FAS=all subjects who took at least 1 dose of study drug and had at least 1 post-baseline measurement. LOCF imputed missing data with any post-baseline visit. Number of subjects with BMI measurements at Baseline and Week 26: inhaled human insulin n=192, insulin glargine n=183.
Measure: Mean (Standard Deviation); unit: kg/m2
Arm/Group | Inhaled Human Insulin | Insulin Glargine
Number analyzed (Participants) | 203 | 189
kg/m2 | 1.22 (1.66) | 0.80 (1.30)
Statistical Analysis 1: Comparison: Inhaled Human Insulin vs Insulin Glargine; Test type: Superiority or Other; p = 0.0053, ANCOVA; Mean Difference (Final Values) = 0.42, 95% CI [0.12 to 0.71]

20. Secondary Outcome: Change From Baseline in Diabetes Treatment Satisfaction Questionnaire-Status, Diabetes Treatment Satisfaction Questionnaire-Change, Diabetes-39, Mental Health Inventory-17, and SF-36 Vitality Domain Questionnaire
Description: Due to cancellation of the EXUBERA program, the collected Patient Reported Outcome (PRO) data, including the Diabetes Treatment Satisfaction Questionnaire-Status, Diabetes Treatment Satisfaction Questionnaire-Change, Diabetes-39, Mental Health Inventory-17, and SF-36 vitality domain questionnaire were not summarized, and no statistical analyses were performed.
Time Frame: Baseline, Week 26
Reporting Status: Not Posted

21. Other Pre Specified Outcome: Change From Baseline in Glycosylated Hemoglobin A1c (HbA1c) at Week 26 for the FAS
Description: HbA1c lab value: Change = value at Week 26 minus value at Baseline.
Time Frame: Baseline, Week 26
Population: FAS=all subjects who took at least 1 dose of study drug and had at least 1 post-baseline measurement. LOCF imputed missing data with any post-baseline visit. Using the FAS yielded supplemental analyses for the primary efficacy endpoint.
Measure: Mean (Standard Deviation); unit: percent
Arm/Group | Inhaled Human Insulin | Insulin Glargine
Number analyzed (Participants) | 203 | 189
percent | -1.91 (1.41) | -1.67 (1.38)
Statistical Analysis 1: Comparison: Inhaled Human Insulin vs Insulin Glargine; [analysis description as in outcome 1, analysis 1]; Test type: Non-Inferiority or Equivalence — The non-inferiority test utilized a one-sided 2.5% level of significance; p < 0.0001, ANCOVA; Mean Difference (Final Values) = -0.27, 95% CI [-0.47 to -0.08] — A CI approach was presented with a two-sided 95% CI of the difference between treatment and control
Statistical Analysis 2: Comparison: Inhaled Human Insulin vs Insulin Glargine; With an established non-inferiority claim, an additional test for superiority was conducted (ie, the margin was 0.0%); Test type: Superiority or Other; p = 0.0062, ANCOVA; Mean Difference (Final Values) = -0.27, 95% CI [-0.47 to -0.08] — The superiority test used a one-sided 2.5% level of significance

ADVERSE EVENTS:
Arm/Group | Inhaled Human Insulin | Insulin Glargine
Serious Adverse Events (participants affected / at risk) | 9 | 4
Other Adverse Events (participants affected / at risk) | 177 | 142
SERIOUS ADVERSE EVENTS; cells are participants affected / at risk:
Term (organ system) | Inhaled Human Insulin | Insulin Glargine
Angina pectoris (Cardiac disorders) | 1/212 | 1/190
Angina unstable (Cardiac disorders) | 1/212 | 0/190
Cardiovascular disorder (Cardiac disorders) | 0/212 | 1/190
Palpitations (Cardiac disorders) | 1/212 | 0/190
Pancreatitis (Gastrointestinal disorders) | 2/212 | 0/190
Chest pain (General disorders) | 1/212 | 0/190
Hepatitis A (Infections and infestations) | 1/212 | 0/190
Sepsis (Infections and infestations) | 0/212 | 1/190
Ankle fracture (Injury, poisoning and procedural complications) | 1/212 | 0/190
Transient ischaemic attack (Nervous system disorders) | 1/212 | 0/190
Nephrolithiasis (Renal and urinary disorders) | 1/212 | 0/190
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 0/212 | 1/190
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected / at risk:
Term (organ system) | Inhaled Human Insulin | Insulin Glargine
Vision blurred (Eye disorders) | 14/212 | 6/190
Diarrhoea (Gastrointestinal disorders) | 12/212 | 8/190
Nausea (Gastrointestinal disorders) | 21/212 | 15/190
Asthenia (General disorders) | 28/212 | 17/190
Fatigue (General disorders) | 13/212 | 11/190
Injection site haematoma (General disorders) | 0/212 | 13/190
Oedema peripheral (General disorders) | 11/212 | 9/190
Influenza (Infections and infestations) | 9/212 | 10/190
Nasopharyngitis (Infections and infestations) | 12/212 | 13/190
Upper respiratory tract infection (Infections and infestations) | 23/212 | 29/190
Weight increased (Investigations) | 17/212 | 9/190
Hypoglycaemia (Metabolism and nutrition disorders) | 144/212 | 83/190
Dizziness (Nervous system disorders) | 40/212 | 29/190
Headache (Nervous system disorders) | 29/212 | 17/190
Tremor (Nervous system disorders) | 67/212 | 43/190
Cough (Respiratory, thoracic and mediastinal disorders) | 18/212 | 6/190
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 35/212 | 21/190

LIMITATIONS AND CAVEATS:
Due to cancellation of the EXUBERA program, the collected Patient Reported Outcome (PRO) data were not summarized, and no statistical analyses were performed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of < 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), < 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.